CLINICAL TRIAL: NCT05516771
Title: Evaluation of a Licensed Double-sensor-heat-flux (DHF) Non-invasive Core Temperature Sensor in Small Children and Toddlers Undergoing Surgery
Status: Completed | Type: Observational
Sponsor: Oliver Kimberger (Other)
Responsible Party: Sponsor-Investigator, Oliver Kimberger, Principal Investigator, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: DHF-TaSC
Record Dates: First submitted 2022-08-21; First posted 2022-08-26 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Hypothermia; Anesthesia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- group 1: toddlers and small children undergoing surgery at a tertiary referral, university-affiliated hospital
  Interventions: Device: Tcore™ system

INTERVENTIONS:
Device: Tcore™ system — The Tcore sensor is a double-sensor-heat-flux (DHF) thermometer and consist of two sensors separated by a known thermal resistance. One side is placed directly at the patient's skin and the other is facing the environment. After some equilibration time the core temperature can then be calculated. The sensors are placed above the eye and the sinus frontalis.
  Intended use The Tcore system is a thermometer intended for non-invasive, continuous measurement of the core body temperature of children from 5 years of age, adolescents, and adults. The Tcore system consists of a sensor and an adapter. The adapter is reusable. The sensor is intended for single use. The Tcore system works in adjusted mode, i.e., the core body temperature is determined by a dual sensor.
  Off-Label/Investigational Use In context of this clinical study the Tcore-system will be investigated outside its approved and intended use, namely in children below the age of five and toddlers.

SUMMARY:
Title: Evaluation of a licensed double-sensor-heat-flux (DHF) non-invasive core temperature sensor in small children and toddlers undergoing surgery.

CI/PS identification code: DHF-TaSC Device Name: Tcore™ system (Tcore-Adapter MP00999 & Tcore-Sensor MP 00989) Manufacturer: Drägerwerk AG & CO KGaA Study design: Prospective, single arm, clinical study

Patients:

* Number: 72
* Age / gender: females and males between 0 and 7 years
* Patients of a tertiary referral, university-affiliated hospital undergoing surgery

Exclusion Criterions:

* Operation site, rash or infection that prevents the application of the heat flux thermometers.
* Patients and/or legal guardians not willing to participate in the trial.
* Patients older than 7 years Setting: ORs of a tertiary referral, university-affiliated hospital. Study variables: measurement triplets measured via two double-sensor-heat-flux (DHF) thermometer the Tcore™ (Dräger, Drägerwerk AG & Co KG, 23558 Lübeck, Germany) one placed on the forehead and one on the upper belly and temperature measured by a rectally placed temperature probe.

DETAILED DESCRIPTION:
Body temperature is important for maintaining normal physiological functions. Inadvertent hypothermia as well as pyrexia are associated with higher morbidity and mortality. Consequently, continuous measurement of body temperature is standard of care at intensive care units (ICUs) and in operation rooms (ORs). The use of core temperature measurements such as pulmonary catheter (gold standard), esophageal or urinary probes is recommended because of higher accuracy than non-invasive measuring methods. The double-sensor-heat-flux (DHF) thermometer the Tcore™ (Dräger, Drägerwerk AG & Co KG, 23558 Lübeck, Germany). The DHF thermometers consist of two sensors separated by a known thermal resistance. One side is placed directly at the patient's skin and the other is facing the environment. After some equilibration time the core temperature can then be calculated. To date no study, exist for the use of the Tcore™ thermometer in children or toddlers. Children are at higher risk for hypothermia and perioperative hypothermia is still common in children.(8) The objective is to find a non-invasive core temperature measurement for children to guide perioperative temperature management.

Primary Objective (Hypothesis):

Evaluation of the accuracy of the licensed double-sensor-heat-flux (DHF) thermometer the Tcore™ (Dräger, Drägerwerk AG & Co KG, 23558 Lübeck, Germany) when used for intraoperative core temperature measurement in small children and toddlers.

The Hypothesis is that each of the two temperature measurements obtained with the Tcore™ (forehead, upper belly) have a high level of agreement(<0.5°C) with the standard of care temperature measurements via rectal temperature probe.

Our primary objective is to investigate the agreement between the two temperature measurements obtained with the Tcore™ (Dräger, Drägerwerk AG & Co KGaA, 23558 Lübeck, Germany) placed on the forehead and the upper belly and temperature measured via a rectally placed Medical Level 1 disposable General Purpose Temperature Probe (Smiths Medical Österreich GmbH, Brunn am Gebirge, Austria). Measure triplets of the two Tcore™ sensors and the rectally placed probe are obtained every 3 minutes for up to 12 consecutive hours or for the duration the patient spends in the OR and the recovery room. If the observed limits of agreement (± 1.96 SD around the mean difference), within which 95% of the differences are expected to fall, are clinically acceptable, the methods are considered to agree. We define deviations of +/-0.5°C, a priori, to be acceptable for the Bland Altman method comparison analysis as was done in previous studies.

Intended use The Tcore system is a thermometer intended for non-invasive, continuous measurement of the core body temperature of children from 5 years of age, adolescents, and adults. The Tcore system consists of a sensor and an adapter. The adapter is reusable. The sensor is intended for single use. The Tcore system works in adjusted mode, i.e., the core body temperature is determined by a dual sensor.

Off-Label/Investigational Use In context of this clinical study the Tcore-system will be investigated outside its approved and intended use, namely in children below the age of five and toddlers.

Descriptive statistics:

* For nominal and ordinal data absolute frequencies and percentages, fraction, rate, and incidence will be calculated, if appropriate.
* Continuous data are described by mean ± standard deviation (SD) in case of approximate normal distribution, or by median, interquartile range otherwise.

Endpoint analysis:

For the primary objective, a scatterplot of differences between Tcore and standard measurements and their mean will be produced for each of the two Tcore measurements in relation to the measurement standard (rectal temperature). If the differences prove to be approximately independent for the observed range of temperatures, limits of agreement will be calculated using the method by Zou (2013).(23) If these limits are contained within the acceptable deviation of +/-0.5°C the respective Tcore measurement method will be considered acceptable. Irrespective of the success of the investigation of agreement the results for both Tcore measurement locations will be reported.

For the secondary objective sensitivity and specificity will be calculated with 95% confidence intervals for each Tcore measurement in relation to the measurement standard.

All study data will be queried from the ICCA and from the database of electronic health records the Vienna General Hospital information management system (AKIM; "Allgemeines Krankenhaus Informationsmanagement") (Siemens AG Österreich, Vienna, Austria). Intellispace Critical Care and Anesthesia. After acquisition, patient data will be anonymized, cleaned, and stored in a study database.

Patient identification will contain name, sex, and birthdate. This data will be documented in an excel sheet, protected with a password. All patients will be given a number for pseudonymization. The verification key will be stored on a separate computer in our laboratory. Only specially authorized persons (Dr. Sebastian Zeiner and Prof. Oliver Kimberger) will have access to the data.

All data will be stored on a password secured computer in the laboratory of our department (Department for Anesthesia) at the Medical University of Vienna.

At any time, medical confidentiality will be fulfilled by all persons involved in this project.

ELIGIBILITY:
Inclusion Criteria:

* 0-7 years
* elective surgical procedures with a procedure time of more than 30 min
* operations for which insertion of a rectal temperature probe is clinically indicated as a routine method, (e.g., operations in regional anaesthesia)

Exclusion Criteria:

* rash or infection that prevents the application of the Heat flux thermometers.
* Fragile forehead skin state;
* known allergy to the probe adhesive or any constituent components
* maxillofacial trauma or lesions
* procedures impeding proper placement of the Tcore™ sensor
* neurologically impaired children with abnormal thermoregulation;
* hemodynamic instability; need for vasoactive medication;
* procedures associated with extended use of abdomino/thoracic rinsing fluids;
* thoracoscopic/thoracotomy procedures;
* malignant hyperthermia or family history of malignant hyperthermia
* patient with fever or infection;
* all conditions that might be judged to abnormally alter skin perfusion
* patients or their legal guardian are not willing to participate in the trial.

Ages: 0 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study population: toddlers and small children undergoing surgery at a tertiary referral, university-affiliated hospital
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02-26 (Actual); Study Completion 2023-02-26 (Actual)

PRIMARY OUTCOMES:
Accuracy of Tcore core temperature measurements | For the duration of Anesthesia and a maximum of 12 hours
  A scatterplot of differences between Tcore and standard measurements of body temperature,limits of agreement will be calculated using the method by Zou (2013).(23)

SECONDARY OUTCOMES:
sensitivity and specificity | For the duration of Anesthesia and a maximum of 12 hours
  For the secondary objective sensitivity and specificity will be calculated with 95% confidence intervals for each Tcore measurement in relation to the measurement standard

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Univercity Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No